CLINICAL TRIAL: NCT00138242
Title: Phase II Trial of Weekly Docetaxel (Taxotere®) and Carboplatin as Initial Chemotherapy for Women With Ovarian Cancer and Similar Malignancies
Brief Title: Docetaxel and Carboplatin in Treating Patients With Ovarian Epithelial, Fallopian Tube, or Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Floyd & Delores Jones Cancer Institute at Virginia Mason Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: VMRC-8837; CDR0000439927 (Registry Identifier: PDQ (Physician Data Query)); AVENTIS-VMRC-8837
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2006-10

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Docetaxel; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: carboplatin
Drug: docetaxel
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel together with carboplatin works in treating patients with ovarian epithelial, fallopian tube, or peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether weekly administration of docetaxel and carboplatin is safer than conventional three-week chemotherapy courses, in terms of reducing the rate of myelosuppression, in patients with stage IC-IV ovarian epithelial, fallopian tube, or peritoneal cavity cancer.

Secondary

* Determine the quality of life of patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine the efficacy of this regimen, in terms of clinical response rate, time to disease progression, and findings at second-look surgery, in these patients.

OUTLINE: Patients receive docetaxel IV and carboplatin IV on days 1, 8, 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients may then undergo optional second-look surgery. After completion of 6 courses of chemotherapy (and second-look surgery, if applicable), patients may receive consolidation and/or salvage therapy at the discretion of the investigator.

Quality of life is assessed at baseline, before each treatment course, at the completion of study treatment, and then annually for 2 years.

After completion of study treatment, patients are followed annually for 2 years.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or peritoneal cavity cancer

  * Stage IC-IV disease
  * No borderline or low malignant potential tumors of any stage
* Underwent initial surgical management, including staging, of early stage disease or surgical debulking of advanced stage disease* NOTE: *Patients may delay surgical debulking, if clinically indicated, until after study entry; these patients may receive several courses of neoadjuvant chemotherapy prior to surgical debulking, but before study entry

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* Meets 1 of the following criteria:

  * Alkaline phosphatase (AP) normal AND AST or ALT ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST or ALT normal

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No peripheral neuropathy > grade 1
* No prior malignancy with a poor prognosis that is at risk of relapse during study participation, as determined by the principal investigator
* No history of severe hypersensitivity reaction to drugs formulated with polysorbate 80

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No concurrent chemotherapy for another malignancy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-12; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Reduction rate of myelosuppression

SECONDARY OUTCOMES:
Quality of life as assessed by the Functional Assessment of Cancer Therapy -Ovarian (FACT-O) questionnaire
Toxicity
Clinical response rate
Findings at second look surgery
Time to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Howard G. Muntz, MD, Principal Investigator — Floyd & Delores Jones Cancer Institute at Virginia Mason Medical Center
Locations (1):
- Floyd & Delores Jones Cancer Institute at Virginia Mason Medical Center, Seattle, Washington, United States